CLINICAL TRIAL: NCT02303808
Title: Effect of Introducing a Positive Expiratory Pressure Device During Inhalation of Hypertonic Saline in Patients With Cystic Fibrosis: a Randomized Crossover Trial.
Brief Title: Positive Expiratory Pressure During Inhalation of Hypertonic Saline in Patients With Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad San Jorge (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: FQ_INH_PEP_01; 239|2012 (Other Grant/Funding Number: SEPAR)
Record Dates: First submitted 2014-11-25; First posted 2014-12-01 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Cystic Fibrosis
Keywords: Hyperosmolar agents; Hypertonic saline; Airway clearance techniques; Positive Expiratory Pressure; Autogenic drainage
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- USUAL CARE (No Intervention): Patients will perform the inhalation of the 7% hypertonic saline (following the gold standard recomendation) during 15 minutes. Right after, patients will perform independently their usual session of autogenic drainage during 30 minutes.
- INHALATION WITH PEP DEVICE (Active Comparator): Patients will perform the inhalation of the 7% hypertonic saline (following the gold standard recomendation) combined with a PEP device (Acapella Duet) during 15 minutes. Right after, patients will perform independently their usual session of autogenic drainage during 30 minutes.
  Interventions: Device: INHALATION WITH PEP DEVICE (Acapella Duet)

INTERVENTIONS:
Device: INHALATION WITH PEP DEVICE (Acapella Duet) — Intervention will be performed during 5 consecutive days. The performance order of both arms will be randomized.
  Arms: INHALATION WITH PEP DEVICE

SUMMARY:
This trial aims to analyze whether the inhalation of hypertonic saline combined with a positive expiratory pressure (PEP) device increases the amount of sputum expectorated during the chest physiotherapy session ( inhalation + bronchial drainage).

DETAILED DESCRIPTION:
All patients will perform two different arms of treatment in a crossover randomization. Each arm of treatment will be applied during 5 consecutive days. The wash-out period will be one week. Before starting the trial all patients will do an inhalation formation.

During the study period the patients' pharmacological treatment remains unchanged

ELIGIBILITY:
Inclusion Criteria:

* Pass the inhalation test
* Chronic sputum production, at least ≥ 10 ml /24h
* Cystic Fibrosis (CF) diagnosed ( established by genotype or sweat sodium>70 mmol/l or sweat chloride of>60 mmol/l)
* Clinically stable at the time of recruitment (defined as no requirement for antibiotics or change in respiratory medication in the preceding 4 weeks)
* Trained in the use of autogenic drainage technique (at least 6 months)
* Inhaling hypertonic saline since at least 6 months
* To be able to provide written, informed consent and perform the protocol and the evaluations

Exclusion Criteria:

* Active massive hemoptysis during the previous 2 months
* Patient in transplantation or retransplantation list
* Patient already participating in another study at the same time

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-12; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Wet sputum production | 45 minutes
  Wet sputum production (ml) during chest physiotherapy session (inhalation + bronchial drainage)

SECONDARY OUTCOMES:
Wet sputum production | 2 hours
  2 hours wet sputum production (ml) after chest physiotherapy session
Wet sputum production | 22 hours
  22 hours wet sputum production (ml) after chest physiotherapy session
Lung function (simply spirometry) | 5 days
  Forced expiratory volume at 1 second, Forced vital capacity, Forced expiratory flow 25-75
Safety and tolerability of session (Pulse-oximetry, heart rate, dyspnea, hemoptysis, cough, throat irritability and saltiness, heart rate) | 45 minutes
  Pulse-oximetry, heart rate, dyspnea, hemoptysis, cough, throat irritability and saltiness, heart rate
Patient's perception (Likert test) | 5 days
  Likert test
Questionnaire | 5 days
  Leicester Cough Questionnaire (LCQ) and Cough and sputum Questionnaire (C&S)

CONTACTS AND LOCATIONS:
Overall Officials: Marta San Miguel, Principal Investigator — Universidad San Jorge
Locations (1):
- Asociación Aragonesa de Fibrosis Quística, Zaragoza, Spain

REFERENCES:
- [Derived] Wark P, McDonald VM, Smith S. Nebulised hypertonic saline for cystic fibrosis. Cochrane Database Syst Rev. 2023 Jun 14;6(6):CD001506. doi: 10.1002/14651858.CD001506.pub5. PMID 37319354
- [Derived] San Miguel-Pagola M, Reychler G, Cebria I Iranzo MA, Gomez-Romero M, Diaz-Gutierrez F, Herrero-Cortina B. Impact of hypertonic saline nebulisation combined with oscillatory positive expiratory pressure on sputum expectoration and related symptoms in cystic fibrosis: a randomised crossover trial. Physiotherapy. 2020 Jun;107:243-251. doi: 10.1016/j.physio.2019.11.001. Epub 2019 Nov 11. PMID 32026826